CLINICAL TRIAL: NCT05522504
Title: Distribution of Immune Cells and Their Subtypes in Peripheral Blood of Gout
Status: Active, not recruiting | Type: Observational
Sponsor: Ai Peng (Other)
Responsible Party: Sponsor-Investigator, Ai Peng, Director of the department of Nephrology, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: SHSY-IEC-4.1/21-246/01
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Gout Flare; Intercritical Gout; Advanced Gout; Asymptomatic Hyperuricemia
Keywords: PBMC monocyte Treg

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- NC: healthy volunteer (Normal control)：(1) aged between 18 and 80 years; (2) The serum UA levels were lower than 420 μmol/L for a man and 360 μmol/L for a woman at least one time during the two clinical tests for the samples collected with 1-week interval; (3) without any clinically diagnostic severe diseases including but not limited to a tumor, diabetes, cardiovascular, renal, nervous, digestive and mental disorders
- AHU: Asymptomatic Hyperuricemia（AHU） were listed as follows: (1) aged between 18 and 80 years; (2) serum levels of UA were both greater than 420 μmol/L for a man and 360 μmol/L for a woman during the two clinical tests for the samples collected with about 1-week interval; (3) without self-reported history of the acute attack of gout; (4) without receiving medical treatment.
- AGA: Acute Gout Attack (AGA) were listed as follows: (1) age between 18 and 80 years; (2) diagnosis with AG at this hospital according to the criteria approved by the ACR Board of Directors and the EULAR Executive Committee in 2015; (3) and not receiving medical treatment 3 weeks prior to the blood collection.
- IG: The intercritical gout (IG) remission criteria for gout patients were listed as follows: (1) age between 18 and 80 years; (2) diagnosis with AG at this hospital according to the criteria approved by the ACR Board of Directors and the EULAR Executive Committee in 2015; (3) remission of clinical manifestations including redness, swelling, heat, and pain at local joint or bursa for at least three months since the last gout flare; (4) normal level (<8.20 mg/L) of C-reactive protein (CRP) at the time of blood collection; (5) without tophi, imaging erosion, or chronic gouty arthritis
- AG: The Advanced gout (AG) criteria for gout patients were listed as follows:(1) age between 18 and 80 years; (2) diagnosis with AG at this hospital according to the criteria approved by the ACR Board of Directors and the EULAR Executive Committee in 2015; (3) remission of clinical manifestations including redness, swelling, heat, and pain at local joint or bursa for at least three months since the last gout flare; (4) normal level (<8.20 mg/L) of C-reactive protein (CRP) at the time of blood collection; (5) with tophi, imaging erosion, or chronic gouty arthritis

SUMMARY:
The purpose of this study is to evaluate whether immune cells and their subtypes in peripheral blood affects the asymptomatic hyperuricemia, gout flare, intercritical gout and advanced gout.

DETAILED DESCRIPTION:
A number of studies have reported that innate immunity cells (such as blood monocytes and neutrophils) play a crucial role in the initiation and amplification of gout flare resulted from MSU deposition in the joint or tissue, leading to release NLRP3 inflammasome-mediated production of bioactive IL-1β. Further investigation demonstrated the role of blood neutrophils might contribute to the resolution of gout flare by forming aggregated neutrophil extracellular traps. Recently, a few in vitro experiments have indicated that adaptive immunity may be involved in mechanisms of gout. However, a global understanding of blood immune responses underlying gout is still unclear. Thus, we want to investigate the relationship between immune cells and their subtypes in peripheral blood and the gout.

ELIGIBILITY:
Inclusion Criteria:

* gout flare:diagnosis with gout flare at this hospital according to the criteria approved by the ACR Board of Directors and the EULAR Executive Committee in 2015
* intercritical gout: remission of gout patients were classified into intercritical gout group without tophi, chronic gouty arthritis, or imaging erosion(All of these gout remission patients underwent dual-energy CT test within one month, and were detected to have MSU crystal deposition in local joints)
* advanced gout: gout remission patients were classified into advanced gout group characterized by tophi, chronic gouty arthritis, or imaging erosion(All of these gout remission patients underwent dual-energy CT test within one month, and were detected to have MSU crystal deposition in local joints)
* asymptomatic hyperuricemia: hyperuricemia in men was defined as SUA ≥ 420 mmol/L without any complications

Exclusion Criteria:

* primary osteoarticular diseases
* unwilling participation in the study
* corticosteroids or indomethacin use in the past 3 months;
* septic arthritis or another joint disease (such as rheumatoid arthritis);
* impaired renal function (creatinine clearance <30 mL/min) and other conditions which may increase the level of blood uric acid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic hyperuricemia Gout flare patients Gout remission patients were classified into intercritical gout group without tophi, chronic gouty arthritis, or imaging erosion, while others were classified into advanced gout group characterized by tophi, chronic gouty arthritis, or imaging erosion.(All of these gout remission patients underwent dual-energy CT test within one month, and were detected to have MSU crystal deposition in local joints) Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
remission of gout | 6 month
  Patients fulfilling all the domains of the 2016 preliminary remission criteria for gout were defined as gout remission group

CONTACTS AND LOCATIONS:
Overall Officials: Ai Peng, MD, PhD, Study Director — Shanghai 10th People's Hospital
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No